CLINICAL TRIAL: NCT07098117
Title: A Randomized, Double-blind, Placebo-controlled Phase I Clinical Trial to Evaluate the Safety and Pharmacokinetic Profile of Single and Multiple Dose Escalation Topical Dermal Administration of SHR0302 Alkali Gel in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHR0302Base-101
Record Dates: First submitted 2025-07-27; First posted 2025-08-01 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Preoperative Sedation of Adults

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 :SHR0302 Base Gel (Experimental)
  Interventions: Drug: SHR0302 Base Gel
- Group2: SHR0302 Base Gel Placebo (Placebo Comparator)
  Interventions: Drug: SHR0302 Base Gel Placebo

INTERVENTIONS:
Drug: SHR0302 Base Gel — Part I: once daily. Part 2:, twice daily.
  Arms: Group 1 :SHR0302 Base Gel
Drug: SHR0302 Base Gel Placebo — Part I: once daily. Part II: twice daily.
  Arms: Group2: SHR0302 Base Gel Placebo

SUMMARY:
This study is divided into two parts, the first part is a single-dose dose escalation trial (SAD) in healthy subjects; The second part is a multiple-dose dose escalation trial (MAD) in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Sign the informed consent form before the trial, fully understand the content, process and possible adverse reactions of the trial, and be able to complete the study according to the requirements of the trial protocol.
2. Must be ≥ 18 years old and ≤ 55 years old on the day of signing the informed consent form, male or female;
3. Male subjects weigh ≥ 50 kg, female subjects weigh ≥ 45 kg, and body mass index (BMI) within the range of 18.0~28.0 kg/m2 (including boundary values);
4. Subjects and their partners have no birth plan, do not donate sperm/eggs, and voluntarily take highly effective contraceptive measures (see Appendix 11 for specific contraceptive measures) from the study period to 6 months (female subjects) or 3 months (male subjects) after dosing, and the serum pregnancy test for female subjects must be negative and non-lactating.

Exclusion Criteria:

1. Those who have had or are currently suffering from any clinically serious diseases such as circulatory system, endocrine system, nervous system, digestive system, respiratory system, blood system, immune system, psychiatric and metabolic abnormalities, or any other diseases that may interfere with the results of the trial in the judgment of the investigator;
2. In the opinion of the investigator, the subject has skin lesions or abnormalities that may affect the evaluation of the study drug administration site, such as dermatitis, tattoos, scars, excessive hair, birthmarks, injuries, uneven skin tone, sunburn, etc.;
3. Subjects have skin diseases that may affect the evaluation at the site of administration, such as vitiligo, eczema, acne, atopic dermatitis, dysplastic moles, or other skin lesions, or a history of skin cancer;
4. Those who have had serious infection, severe trauma or major surgical surgery within 6 months before screening; Those who plan to undergo surgery during the trial and within 2 weeks of the end;
5. Positive hepatitis B virus surface antigen (HBsAg), human immunodeficiency virus antibody (HIV-Ab), Treponema pallidum antibody, and hepatitis C virus antibody (HCV-Ab) during the screening period;
6. Estimated glomerular filtration rate (eGFR) calculated by the Dietary Modification for Nephrology (MDRD) formula (see Appendix 2) < 90 mL/min/1.73 m² at screening, or serum creatinine exceeding the normal range, and judged by the investigator to be clinically significant and not suitable for participation in this investigator;
7. Suspected allergy to the test drug or any ingredient in the test drug;
8. Abnormal vital signs, physical examination, laboratory tests (blood routine, urine routine, blood biochemistry, coagulation function), chest stereotype, abdominal ultrasound and 12-lead electrocardiogram at screening and judged by the investigator to be unsuitable for participation in this study;
9. Screening or baseline 12-lead ECG QTcF>450 ms and abnormal clinically significant as judged by the investigator;
10. Screening or baseline systolic blood pressure ≥ 140 mmHg or < 90 mmHg; Diastolic blood pressure ≥ 90 mmHg or < 60 mmHg, and abnormal clinically significant as judged by the investigator;
11. Subjects who have a test result of 1.5 times the upper limit of normal (ULN) > any of the test results of alanine aminotransferase (ALT), or aspartate aminotransferase (AST), or total bilirubin (TBIL) at screening or baseline;
12. Those who have used any drugs within 2 weeks before the first use of the investigational drug or those who have used the drug for less than 5 half-lives (whichever is longer), and those who plan to use any other drugs during the study, including prescription drugs, over-the-counter drugs, Chinese herbal medicines and food supplements (except oral contraceptives), etc.;
13. The subject has any conditions or diseases that affect the absorption, metabolism and/or excretion of the trial drug as judged by the investigator;
14. Those who have participated in any clinical trial of any drug or medical device within 3 months before screening, or who are within 5 half-lives of the drug before screening (if the 5 half-lives exceed 3 months, whichever is longer); Participants in clinical trials are defined as: informed consent from clinical trials, and have used investigational drugs (including placebos) or experimental medical devices;
15. Those who have received live (attenuated) vaccines 1 month before screening or plan to receive live (attenuated) vaccines during the trial;
16. Total blood donation or blood loss ≥ 200 mL within 1 month prior to screening, or total blood donation or blood loss ≥ 400 mL within 3 months prior to screening; or those who have received blood transfusion within 2 months; or those who have difficulty in venous blood collection, or whose physical condition cannot bear intensive blood collection;
17. Those who have a history of smoking in the 3 months before screening (smoking > 5 cigarettes per day);
18. Alcoholics (drinking 14 units of alcohol per week [1 unit = 285 mL of beer, or 25 mL of spirits, or 100 mL of wine]) or positive alcohol breath test at baseline within 3 months prior to screening;
19. Those who cannot abstain from smoking, alcohol and caffeinated food or beverages 2 days before and during the study of the investigational drug; and those who have special requirements for diet and cannot comply with the unified diet;
20. Those with a history of drug abuse, drug dependence, or positive drug screen at baseline;
21. Pregnant or lactating women, pregnancy is defined as female status after pregnancy to before termination of pregnancy and positive blood β-HCG test at screening;
22. Have any situation that may cause the subject to be unable to complete this study or pose obvious risks to the subject or other factors that reduce the possibility of enrollment (such as frailty, mental illness, etc.);
23. Researchers and relevant staff of the research center or other people directly involved in the implementation of the program.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2024-06-19 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Part 1, Skin local tolerability was assessed as moderate and above incidence, adverse events | 8days
Part 2, Skin local tolerability was assessed as moderate and above incidence, adverse events | 2weeks

CONTACTS AND LOCATIONS:
Locations (1):
- The First Hospital of Jilin University, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: Undecided